CLINICAL TRIAL: NCT06537245
Title: Does Application Time Influence the Effect of Massage on Pain and Performance? A Crossover Randomized Controlled Tria
Brief Title: Does Application Time Influence the Effect of Massage on Pain and Performance?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual do Norte do Parana (Other)
Responsible Party: Principal Investigator, Jéssica Kirsch Micheletti, Principal Investigator, Universidade Estadual do Norte do Parana
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: UNorteParana
Record Dates: First submitted 2024-02-20; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Health, Subjective
Keywords: Massage; Recovery of Function; Muscle Strength
MeSH Terms: interventions — Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 minutes massage group (Experimental): The anatomical location chosen for applying the massage was the anterior part of the thigh (muscular quadriceps femoris), due to the effort required by the stress protocol.
  The participant was placed in the supine position and the massage was performed on the dominant limb (DOM) and the non-dominant limb (ÑDOM). The techniques used were: superficial and deep sliding, which is presented in two intensities, moderate or intense, with gradual increase. Intensity grading was controlled through participant self-reports. The massage was performed in the direction of the muscle fibers, from distal to proximal and following the lymphatic flow.
  The massage had the following rhythm: 1 second of sliding and 1 second to return the hand to the initial position, totaling 2 seconds of sliding. The rhythm of the massage was controlled by an electronic metronome that was used only by the therapists during the technique.
  Interventions: Other: Massage
- 10 minutes massage group (Experimental): The anatomical location chosen for applying the massage was the anterior part of the thigh (muscular quadriceps femoris), due to the effort required by the stress protocol.
  The participant was placed in the supine position and the massage was performed on the dominant limb (DOM) and the non-dominant limb (ÑDOM). The techniques used were: superficial and deep sliding, which is presented in two intensities, moderate or intense, with gradual increase. Intensity grading was controlled through participant self-reports. The massage was performed in the direction of the muscle fibers, from distal to proximal and following the lymphatic flow.
  The massage had the following rhythm: 1 second of sliding and 1 second to return the hand to the initial position, totaling 2 seconds of sliding. The rhythm of the massage was controlled by an electronic metronome that was used only by the therapists during the technique.
  Interventions: Other: Massage

INTERVENTIONS:
Other: Massage — Massage was applied in the both quads during 5 or 10 minutes, with differents pressures.

SUMMARY:
Introduction: The massage technique is widely used for post-exercise recovery, however, there is still a gap regarding the ideal dosage in relation to the duration of its application. Objective: To analyze the influence of massage when applied at different times on the dominant (DOM) and non dominant (ÑDOM) quadriceps muscles and clinical variables. Methods: Study carried out with 11 men aged 21.5(2.1) years, in a two-week crossover design. Participants performed a jumping protocol followed by manual massage for 5 (G1) or 10 (G2) minutes. Assessments included strength testing, pain scale (VAS), perception of recovery and vital sign measurements up to one hour post-massage. Analysis onducted in SPSS, ANOVA was performed (with Bonferroni test, when necessary), providing effect sizes (p<0.05).

DETAILED DESCRIPTION:
The massage technique is widely used for post-exercise recovery, however, there is still a gap regarding the ideal dosage in relation to the duration of its application. The objective was to analyze the influence of massage when applied at different times with the participation of 11 men, in a two-week crossover design. Participants performed a jumping protocol followed by manual massage for 5 (G1) or 10 (G2) minutes. Assessments included strength testing, pain scale (VAS), perception of recovery and vital sign measurements up to one hour post-massage.

ELIGIBILITY:
IInclusion Criteria:

* Students
* Mens
* Aged 18 to 35 years
* Healthy (self-report) regularly enrolled in the Physiotherapy course at the Northern Paraná State University (UENP), from the 1st to the 5th year
* Who have not undergone
* Surgery in the last spine and lower limbs and were instructed not to perform any physical activity in the last 24 hours before the test.

Exclusion Criteria:

* People who are not enrolled in the Physiotherapy course at the State University of Northern Paraná
* Are not in good health
* Have undergone surgery on the lower limbs within a period of 12 months
* Have practiced physical activity in the last 24 hours

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 11 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Muscle Strenght. | Pre stress protocol and 40 minutes post stress protocol.
  Isokinetic Device.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Micheletti, Study Director — UNorteParaná
Locations (1):
- UNorteParana, Jacarezinho, PR - Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No